CLINICAL TRIAL: NCT00058058
Title: MRI Evaluation Of The Contralateral Breast In Women With Recent Diagnosis Of Breast Cancer
Brief Title: Magnetic Resonance Imaging in Women Recently Diagnosed With Unilateral Breast Cancer
Acronym: ACRIN-6667
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000285698; ACRIN-6667 (Other: American College of Radiology Imaging Network); U01CA079778 (NIH); U01CA080098 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Contralateral Breast Cancer
Keywords: ductal breast carcinoma in situ; invasive ductal breast carcinoma; invasive lobular breast carcinoma; breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; Magnetic resonance imaging; MRI
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Breast Carcinoma In Situ | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Evaluation of Contralateral Breast (Experimental): The cohort is a distinct population of women at high risk for breast carcinoma: women with a recent (within 60 days) personal diagnosis of breast cancer who will have MRI to evaluate the contralateral breast.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Breast contralateral to the breast diagnosed with cancer was scanned prior to initiation of chemotherapy and within 90 days of a negative mammogram of the study breast. A recent (within 90 days) negative or benign mammogram (defined by final BI RADS category 1 or 2) and negative or benign clinical breast exam of the study breast were required for entry into the study.
  Other Names: magnetic resonance imaging

SUMMARY:
RATIONALE: Diagnostic procedures such as magnetic resonance imaging (MRI) may improve the ability to detect cancer in the unaffected breast of women recently diagnosed with unilateral breast cancer.

PURPOSE: Diagnostic trial to determine the effectiveness of MRI in evaluating the unaffected breast of women recently diagnosed with unilateral breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the diagnostic yield of magnetic resonance imaging (MRI) in evaluating the contralateral breast of women with a recent unilateral diagnosis of breast cancer and a negative contralateral mammogram and clinical breast exam.
* Determine the sensitivity, specificity, positive predictive value for both call backs for additional imaging and biopsy recommendations, and receiver operating characteristic curves of MRI in evaluating these patients.
* Determine the effect of the following patient-related factors: age (50 years old and over vs less than 50 years old), breast parenchymal density (fatty vs non fatty breast), and tumor histology (invasive lobular vs invasive ductal, invasive vs in situ) on the performance of MRI (cancer yield, sensitivity, specificity, and PPV).

OUTLINE: This is a multicenter study.

Patients receive gadopentetate dimeglumine IV and then undergo magnetic resonance imaging of the contralateral breast.

Patients are followed at 12-18 and 24-30 months.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Recently confirmed unilateral ductal carcinoma in situ or invasive cancer of the breast

  * Confirmed by biopsy or fine needle aspiration (FNA) within the past 60 days
* Negative or benign mammogram (BI-RADS assessment 1 or 2) and negative or benign clinical breast exam of the contralateral breast within the past 90 days
* Prior biopsy of the contralateral breast (including FNA) is allowed provided it was performed at least 6 months prior to study entry
* Prior magnetic resonance exam of the contralateral breast is allowed provided it was performed at least 1 year prior to study entry
* No remote history of breast cancer
* No new breast symptoms within the past 60 days for which further evaluation is recommended
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No pacemaker
* No magnetic aneurysm clips

Other

* Not pregnant
* No implanted magnetic device
* No severe claustrophobia
* No other contraindications to MRI
* No psychiatric, psychological, or other condition that would preclude informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 6 months since prior anticancer chemotherapy

Endocrine therapy

* No concurrent therapeutic hormonal therapy, tamoxifen, or aromatase inhibitors (preventive therapy allowed)

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2006-08-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Lehman, MD, PhD, Study Chair — Seattle Cancer Care Alliance
Locations (21):
- United States (19):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Porter Adventist Hospital, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada
- Universitaetsklinikum Bonn, Bonn, Germany

REFERENCES:
- [Result] DeMartini WB, Hanna L, Gatsonis C, Mahoney MC, Lehman CD. Evaluation of tissue sampling methods used for MRI-detected contralateral breast lesions in the American College of Radiology Imaging Network 6667 trial. AJR Am J Roentgenol. 2012 Sep;199(3):W386-91. doi: 10.2214/AJR.11.7000. PMID 22915431
- [Result] Weinstein SP, Hanna LG, Gatsonis C, Schnall MD, Rosen MA, Lehman CD. Frequency of malignancy seen in probably benign lesions at contrast-enhanced breast MR imaging: findings from ACRIN 6667. Radiology. 2010 Jun;255(3):731-7. doi: 10.1148/radiol.10081712. PMID 20501712
- [Result] Lehman CD, Gatsonis C, Kuhl CK, Hendrick RE, Pisano ED, Hanna L, Peacock S, Smazal SF, Maki DD, Julian TB, DePeri ER, Bluemke DA, Schnall MD; ACRIN Trial 6667 Investigators Group. MRI evaluation of the contralateral breast in women with recently diagnosed breast cancer. N Engl J Med. 2007 Mar 29;356(13):1295-303. doi: 10.1056/NEJMoa065447. Epub 2007 Mar 28. PMID 17392300
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data includes information on 1007 participants enrolled between April 1, 2003 and June 10, 2004 at 25 centers for data collected through August 8, 2006.
Pre-assignment Details: Patients were not imaged by MRI if they did not meet eligibility criteria, withdrew, or were otherwise unable to be scanned (claustrophobic, too large for scanner, illness, etc.)
Period: Overall Study
Arm/Group | MRI Evaluation of Contralateral Breast
Started (Enrolled) | 1007
Completed (Completed MRI) | 969
Not Completed | 38
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible | 20
Not completed — Claustrophobic | 5
Not completed — technical issues | 6
Not completed — Poor positioning, illness,pain | 3

BASELINE CHARACTERISTICS:
Arm/Group | MRI Evaluation of Contralateral Breast
Number analyzed (Participants) | 969
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 969
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 925
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2
  Asian | 23
  Black or African American | 48
  Native Hawaiian Pacific Islander | 2
  White | 887
  Unknown | 14

OUTCOME MEASURES:

1. Primary Outcome: MRI Diagnostic Yield of Cancers in the Contralateral Breast
Description: To assess the diagnostic yield of magnetic resonance imaging (MRI) in evaluating the contralateral breast of women with a recent unilateral diagnosis of breast cancer and a negative contralateral mammogram and clinical breast exam.
  the "Test" status was defined based on combinations of the following 4 factors:
  1. The initial BI-RADs: from the MRI of the contralateral breast
  2. The final BI-RADs: determined after all subsequent work-up and follow-up within 365 from the initial MRI (an explicit recommendation for biopsy always resulted in a final BI-RADs of 4).
  3. Subsequent work-up includes all procedures resultant from an Initial MRI finding (generally triggered by a BI-RADs 0 or 3) within 365 from the initial MRI
  4. Whether or not biopsy procedure (Bx) were performed on the contralateral (Study) breast within 365 from the initial MRI
Time Frame: within 90 days of a negative mammogram of the study breast
Population: All eligible participants with an analyzable MRI
Measure: Count of Participants; unit: Participants
Groups:
- Reference Standard Positive (RS+): Reference Standard Positive indicates a breast cancer diagnosed in the contralateral (study) breast. Participants who received a diagnosis of ductal carcinoma in situ or any invasive breast cancer as a result of a biopsy or surgery that was performed within 365 days of the initial MRI scan were considered positive for cancer. Participants were considered positive only on the basis of positive tissue diagnosis.
- Reference Standard Negative (RS-): Women with no diagnosis of cancer during the year after their enrollment were considered negative. All cases for whom no tissue diagnosis of cancer was reported during the 365 days following the initial MRI were considered negative, regardless of whether any additional imaging had been performed.
Arm/Group | Reference Standard Positive (RS+) | Reference Standard Negative (RS-)
Number analyzed (Participants) | 33 | 936
Participants
  Test + (Final BI-RAD 0, 4, 5): Test Positive (T+) | 30 | 114
  Test + (Final BI-RAD 0, 4, 5): Test Negative (T-) | 3 | 822
  Test + (Initial MRI BI-RAD 4, 5/work-up): Test Positive (T+) | 30 | 105
  Test + (Initial MRI BI-RAD 4, 5/work-up): Test Negative (T-) | 3 | 831
  Test + (Initial MRI BI-RAD 4, 5/work-up/comp bx): Test Positive (T+) | 30 | 91
  Test + (Initial MRI BI-RAD 4, 5/work-up/comp bx): Test Negative (T-) | 3 | 845
  Test + (Initial MRI BI-RAD 0, 4, 5): Test Positive (T+) | 30 | 143
  Test + (Initial MRI BI-RAD 0, 4, 5): Test Negative (T-) | 3 | 793
  Test + (Initial MRI BI-RAD 0, 3, 4, 5): Test Positive (T+) | 31 | 247
  Test + (Initial MRI BI-RAD 0, 3, 4, 5): Test Negative (T-) | 2 | 689
  Test + (Initial MRI BI-RAD 0, 3, 4, 5/work-up)".: Test Positive (T+) | 31 | 145
  Test + (Initial MRI BI-RAD 0, 3, 4, 5/work-up)".: Test Negative (T-) | 2 | 791
Statistical Analysis 1: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 0, 4 or 5 based on Final BI-RADS; Test type: Other — Estimation of diagnostic yield; Binomial proportion = 0.031, 95% CI 2-sided [0.020 to 0.042], Standard Error of Mean 0.006
Statistical Analysis 2: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 4 or 5 based on initial MRI and subsequent work-up; Test type: Other; Binomial Proportion = 0.031, 95% CI 2-sided [0.021 to 0.044], Standard Error of Mean 0.006
Statistical Analysis 3: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 4 or 5 based on initial MRI and subsequent work-up and a completed biopsy procedure; Test type: Other; Binomial Proportion = 0.031, 95% CI 2-sided [0.020 to 0.042], Standard Error of Mean 0.006
Statistical Analysis 4: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 0, 4 or 5 on the initial MRI scan; Test type: Other; Binomial proportion = 0.031, 95% CI 2-sided [0.020 to 0.042], Standard Error of Mean 0.006
Statistical Analysis 5: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 0, 3, 4 or 5 on the initial MRI scan; Test type: Other; Binomial Proportion = 0.032, 95% CI 2-sided [0.021 to 0.043], Standard Error of Mean 0.006
Statistical Analysis 6: Comparison: Reference Standard Positive (RS+); Diagnostic Yield is defined as the likelihood that a test or procedure will provide the information needed to establish a diagnosis. For this analysis, a Positive Test is defined as a score of BI-RADS 0, 3, 4 or 5 based on initial MRI and subsequent work-up; Test type: Other; Binomial Proportion = 0.032, 95% CI 2-sided [0.021 to 0.043], Standard Error of Mean 0.006

2. Secondary Outcome: MRI Detection of Cancer in the Contralateral Breast for the Estimation of Diagnostic Accuracy
Description: Accuracy values (Sensitivity, Specificity, Positive Predicative Value (PPV), Negative Predictive Value (NPV), Diagnostic Yield, and Area Under the Curve (AUC)) of MRI in evaluating the contralateral breast of women with recent personal diagnosis of breast cancer will be determine from the reference standard (a diagnosed cancer in the study breast) and the Test result defined as either the Probability of malignancy from the initial MRI interpretation (for AUC) or the "Final BI-RADs", where the final BI-RADS is defined as the BI-RADS assigned after all subsequent work-up and follow-up within 365 from the initial MRI are complete (an explicit recommendation for biopsy always results in a final BI-RADs of 4).
Time Frame: within 90 days of a negative mammogram of the study breast
Population: All eligible participants with an analyzable MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Standard Positive (RS+) | Reference Standard Negative (RS-)
Number analyzed (Participants) | 33 | 936
Participants
  Test + (Final BI-RAD 0, 4, 5) | 30 | 114
  Test - (Final BI-RAD 1,2,3) | 3 | 822
Statistical Analysis 1: Comparison: Reference Standard Positive (RS+); Sensitivity estimate - estimates the P(T+|D+) where the MRI within 90 days of a negative mammogram is the test (T) and cancer in the contralateral breast is the Disease status(D); Test type: Other; Binomial Proportion = 0.9091, 95% CI 2-sided [0.7567 to 0.9809], Standard Error of Mean 0.05004
Statistical Analysis 2: Comparison: Reference Standard Negative (RS-); Specificity - estimates the P(T-|D-) of MRI where the MRI within 90 days of a negative mammogram is the test (T) and cancer in the contralateral breast is the Disease status(D); Test type: Other; Binomial Proportion = .8782, 95% CI 2-sided [0.8555 to 0.8985], Standard Error of Mean 0.0107
Statistical Analysis 3: Comparison: Reference Standard Positive (RS+) vs Reference Standard Negative (RS-); PPV estimate - estimates the P(D+|T+), where the MRI within 90 days of a negative mammogram is the test (T) and cancer in the contralateral breast is the Disease status(D); Test type: Other; Binomial Proportion = .2083, 95% CI 2-sided [0.1452 to 0.2839], Standard Error of Mean 0.0338
Statistical Analysis 4: Comparison: Reference Standard Positive (RS+) vs Reference Standard Negative (RS-); B. NPV Analysis for ALL Cases in Analysis Set NPV estimate - estimates the P(D-|T-), where the MRI within 90 days of a negative mammogram is the test (T) and cancer in the contralateral breast is the Disease status(D); Test type: Other; Binomial Proportion = 0.9964, 95% CI 2-sided [0.9894 to 0.9993], Standard Error of Mean 0.0021
Statistical Analysis 5: Comparison: Reference Standard Positive (RS+) vs Reference Standard Negative (RS-); B. Diagnostic Yield for ALL Cases in Analysis Set Diagnostic Yield - estimates the likelihood that the MRI within 90 days of a negative mammogram will provide the information needed to establish a diagnosis; Test type: Other; Binomial Proportion = 0.0310, 95% CI 2-sided [0.021 to 0.044], Standard Error of Mean 0.00556

3. Secondary Outcome: AUC as a Measure of the Accuracy of MRI for the Detection of Cancer in the Contralateral Breast
Description: Area Under the Curve (AUC) of MRI in evaluating the contralateral breast of women with recent personal diagnosis of breast cancer will be determine from the reference standard (a diagnosed cancer in the study breast) and the Test result defined as the Probability of malignancy from the initial MRI interpretation.
Time Frame: within 90 days of a negative mammogram of the study breast
Population: All eligible participants with an analyzable MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Standard Positive (RS+) | Reference Standard Negative (RS-)
Number analyzed (Participants) | 33 | 936
Participants
  1: Definitely not malignant | 2 | 565
  2: Probably not malignant | 2 | 256
  3: Possibly malignant | 10 | 92
  4: Probably malignant | 15 | 21
  5: Definitely malignant | 4 | 2
Statistical Analysis 1: Comparison: Reference Standard Positive (RS+) vs Reference Standard Negative (RS-); ROC analysis - estimates the accuracy of MRI within 90 days of a negative mammogram to detect cancer in the contralateral breast; Test type: Other; ROC analysis = 0.9355, 95% CI 2-sided [0.8956 to 0.9753] — exact CI

ADVERSE EVENTS:
Time Frame: 30 DAYS POST Intervention
Arm/Group | MRI Evaluation of Contralateral Breast
All-Cause Mortality (participants affected / at risk) | 0/1007
Serious Adverse Events (participants affected / at risk) | 0/1007
Other Adverse Events (participants affected / at risk) | 0/1007

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No